CLINICAL TRIAL: NCT05022199
Title: Use of SPY Fluorescent Angiography to Reduce Ureteroenteric Stricture Rate Following Urinary Diversion
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Tracey Krupski, MD, Associate Professor, Department of Urology, University of Virginia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSR200414
Record Dates: First submitted 2021-08-23; First posted 2021-08-26 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Ureteral Obstruction; Stricture Ureter
MeSH Terms: conditions — Ureteral Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Study Arm: SPY fluorescent angiography (Experimental)
  Interventions: Device: SPY fluorescent angiography
- Historic Control Arm: Urinary diversion without the use of SPY (No Intervention): This arm consists of 215 historic controls who have undergone urinary diversion at UVA from 2015-2020 without the use of SPY fluorescent angiography

INTERVENTIONS:
Device: SPY fluorescent angiography — This group has had SPY fluorescent angiography used intraoperatively during urinary diversion. To be compared with historic controls who did not.
  Arms: Study Arm: SPY fluorescent angiography

SUMMARY:
Ureteroenteric anastomotic stricture is a well-known complication of urinary diversion which occurs in 4-25% of patients. Recent study has yielded that radiation is a significant risk factor for development of ureteroenteric stricture. The goal of this study is to determine whether intraoperative use of SPY fluorescent angiography during urinary diversion reduces rate of ureteroenteric stricture.

This study will include 215 patients who have undergone urinary diversion over the past 5 years as historic controls and compare ureteroenteric stricture rates to a prospective cohort of patients in whom intraoperative SPY fluorescent angiography was used at the time of urinary diversion to assess the anastomotic perfusion. This will include injection of ICG intravenously as well as utilization of the SPY device to assess ureteral perfusion before and after ureteroenteric anastomosis. Based on power analysis, this study will require approximately 50 patients in our prospective group to detect a clinically significant difference of 5% between groups. Data analysis plan includes the use of chi square test for comparison of stricture rates between groups. Clinical outcomes will be followed prospectively, with no amendment to standard follow-up per physician.

DETAILED DESCRIPTION:
Ureteroenteric anastomotic stricture is a well-known complication of urinary diversion which occurs in 4-25% of patients. Strictures present clinically with flank pain, decreased renal function, pyelonephritis or may be asymptomatic and diagnosed incidentally with progressive hydronephrosis and renal impairment. Strictures are a cause of significant morbidity and health care expenditure, as treatment necessitates procedural intervention and often several inpatient admissions. Numerous studies have sought to identify risk factors for development of ureteroenteric strictures as well as opportunities for technical approaches to reduce stricture risk. Studies have demonstrated that Clavien-Dindo ≥ 3 complication and BMI were associated with higher risk of stricture.

Ischemia of the anastomosis related to the tenuous ureteral blood supply is implicated in the formation of ureteroenteric stricture. Basic science and animal data have established the detrimental impact of radiation therapy on microvasculature. Radiation induced ureteral ischemia in conjunction with periureteral fibrosis make preservation of distal ureteral blood supply during urinary diversion tenuous and challenging. This is especially of concern in patients requiring pelvic exenteration for colorectal or gynecological malignancy, which often necessitate radiation therapy prior to surgical intervention. Radiation history is also an important contributor commonly in patients undergoing benign diversion for radiation cystitis.

Several groups have tested whether varied surgical methods may offer risk reduction. Surgical anastomotic approach has not significantly impacted ureteroenteric stricture rate. However, a more recent study suggests that intracorporeal diversion confers a higher risk of ureteroenteric stricture. The gold standard for treatment of ureteroenteric stricture is open repair with ureteral reimplantation. Open surgical repair has success of 92-100%, while endoscopic management has success of 30-50%.

A recent study demonstrated that through the use of indocyanine green (ICG) fluorescent angiography while performing urinary diversion using the DaVinci robotic system, that they were able to reduce stricture rates from 10.6% to 0%. Use of this technology allows the surgeon to evaluate the vascular supply to the ureter as well as the newly created ureteroenteric anastomosis. This significant reduction in complications has tremendous implications for improvement in patient care and reduction of morbidity. Many patients are not candidates for robotic urinary diversion and thus undergo open surgery. Fluorescent angiography has also shown promise for decreasing ureteroenteric stricture rate in open surgery.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing open urinary diversion

Exclusion Criteria:

* Inability to provide informed consent
* Robotic-assisted urinary diversion
* Pregnant Women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of Ureteroenteric Stricture | 1.5 years

SECONDARY OUTCOMES:
90 day postoperative readmission | 90 days
Rate of hydronephrosis, pyelonephritis, or renal impairment | 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shen JK, Jamnagerwalla J, Yuh BE, Bassett MR, Chenam A, Warner JN, Zhumkhawala A, Yamzon JL, Whelan C, Ruel NH, Lau CS, Chan KG. Real-time indocyanine green angiography with the SPY fluorescence imaging platform decreases benign ureteroenteric strictures in urinary diversions performed during radical cystectomy. Ther Adv Urol. 2019 Apr 4;11:1756287219839631. doi: 10.1177/1756287219839631. eCollection 2019 Jan-Dec. PMID 31057669
- [Background] Ahmadi N, Ashrafi AN, Hartman N, Shakir A, Cacciamani GE, Freitas D, Rajarubendra N, Fay C, Berger A, Desai MM, Gill IS, Aron M. Use of indocyanine green to minimise uretero-enteric strictures after robotic radical cystectomy. BJU Int. 2019 Aug;124(2):302-307. doi: 10.1111/bju.14733. Epub 2019 Apr 11. PMID 30815976
- [Derived] Yeaman C, Ignozzi G, Kazeem A, Isharwal S, Krupski TL, Culp SH. Impact of SPY Fluorescence Angiography on Incidence of Ureteroenteric Stricture After Urinary Diversion. J Urol. 2024 Dec;212(6):844-850. doi: 10.1097/JU.0000000000004198. Epub 2024 Aug 20. PMID 39162209